CLINICAL TRIAL: NCT07370415
Title: Comparison of Ultrasound-Guided Modified Thoracolumbar Interfascial Plane Block Versus Quadro-Iliac Plane Block for Postoperative Analgesia After Lumbar Instrumentation Surgery
Brief Title: mTLIP vs QIPB for Postoperative Analgesia After Lumbar Instrumentation Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Merih Yıldız Eglen, principal investigator, MD, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BursaCity Hos 3
Record Dates: First submitted 2026-01-12; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative
Keywords: Lumbar instrumentation surgery; Postoperative Pain; Modified thoracolumbar interfascial plane block; Quadro-iliac plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Thoracolumbar Interfascial Plane Block (mTLIP) Group (Experimental): Participants in this group will receive a bilateral ultrasound-guided modified thoracolumbar interfascial plane block (mTLIP) performed at the end of lumbar instrumentation surgery while in the prone position. Under sterile conditions, the ultrasound probe will be placed in the parasagittal plane at the midpoint of the surgical incision, taking into account the operated lumbar levels. The paraspinal muscles will be identified, and using an in-plane technique, the needle will be advanced into the interfascial plane between the longissimus and iliocostalis muscles. After confirmation of correct needle placement with saline, 20 mL of 0.25% bupivacaine will be injected on each side. The block will be performed bilaterally, with a total volume of 40 mL of 0.25% bupivacaine.
  Interventions: Procedure: Modified Thoracolumbar Interfascial Plane Block (mTLIP)
- Quadro-Iliac Plane Block (QIPB) Group (Experimental): Participants in this group will receive a bilateral ultrasound-guided quadro-iliac plane block (QIPB) performed at the end of lumbar instrumentation surgery while in the prone position. Under sterile conditions, a convex ultrasound probe will be placed at the point where the quadratus lumborum muscle attaches to the iliac crest. The erector spinae and quadratus lumborum muscles will be identified, and correct needle placement will be confirmed with saline injection. Subsequently, 20 mL of 0.25% bupivacaine will be injected on each side, with visualization of local anesthetic spread between the erector spinae and quadratus lumborum muscles. The block will be performed bilaterally, with a total volume of 40 mL of 0.25% bupivacaine.
  Interventions: Procedure: Quadro-Iliac Plane Block (QIPB):

INTERVENTIONS:
Procedure: Modified Thoracolumbar Interfascial Plane Block (mTLIP) — An ultrasound-guided bilateral fascial plane block in which local anesthetic is injected into the interfascial plane between the longissimus and iliocostalis muscles at the operated lumbar levels. The block is performed under sterile conditions at the end of surgery using 0.25% bupivacaine (20 mL per side; total volume 40 mL).
  Arms: Modified Thoracolumbar Interfascial Plane Block (mTLIP) Group
Procedure: Quadro-Iliac Plane Block (QIPB): — An ultrasound-guided bilateral fascial plane block in which local anesthetic is injected at the point where the quadratus lumborum muscle attaches to the iliac crest, allowing spread between the erector spinae and quadratus lumborum muscles. The block is performed under sterile conditions at the end of surgery using 0.25% bupivacaine (20 mL per side; total volume 40 mL).
  Arms: Quadro-Iliac Plane Block (QIPB) Group

SUMMARY:
Lumbar instrumentation surgery is associated with severe postoperative pain due to extensive tissue dissection and prolonged muscle retraction during the procedure. Inadequate postoperative pain control may result in delayed mobilization, increased cardiopulmonary complications, and prolonged hospital stay. Ultrasound-guided regional analgesia techniques are increasingly used to improve postoperative pain management after lumbar spine surgery. The thoracolumbar interfascial plane (TLIP) block has been shown to provide effective analgesia for lumbar instrumentation surgery, and its modified technique (mTLIP) has been reported to enhance postoperative pain control. The quadro-iliac plane (QIP) block is a newly described fascial plane block with promising results in lumbar spine surgery. This randomized controlled trial aims to compare the postoperative analgesic effectiveness of the modified thoracolumbar interfascial plane block and the quadro-iliac plane block in patients undergoing lumbar instrumentation surgery.

DETAILED DESCRIPTION:
Lumbar instrumentation surgery is commonly associated with moderate-to-severe postoperative pain due to extensive tissue dissection and prolonged muscle retraction. Inadequate pain control may lead to delayed mobilization, increased cardiopulmonary complications, and prolonged hospital stay.

Ultrasound-guided regional analgesia techniques, particularly fascial plane blocks, are increasingly used as part of multimodal analgesia in lumbar spine surgery. The thoracolumbar interfascial plane (TLIP) block is an established technique that provides effective analgesia and has been modified to improve its clinical application, resulting in the modified thoracolumbar interfascial plane (mTLIP) block. Previous studies have demonstrated the effectiveness of mTLIP for postoperative analgesia after lumbar instrumentation surgery.

The quadro-iliac plane block (QIPB) is a recently described ultrasound-guided fascial plane block. Early reports suggest that QIPB may provide effective analgesia in lumbar spine procedures; however, comparative evidence with established techniques remains limited.

This prospective randomized controlled trial aims to compare bilateral ultrasound-guided mTLIP and QIPB performed at the end of surgery in patients undergoing elective lumbar instrumentation surgery under general anesthesia, to evaluate whether QIPB can be considered a safe and effective alternative to mTLIP for postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Classified as American Society of Anesthesiologists physical status I-III
* Scheduled for elective lumbar instrumentation surgery under general anesthesia
* Provision of written informed consent

Exclusion Criteria:

* Use of anticoagulant medications or presence of bleeding diathesis
* Known allergy or hypersensitivity to local anesthetics or opioid drugs
* Infection at the planned block site
* Alcohol or drug dependence
* Cognitive impairment preventing reliable pain assessment
* Pregnancy or lactation
* History of previous lumbar spine surgery
* Diabetes mellitus
* Renal or hepatic insufficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative 48-Hour PCA Opioid Consumption | Postoperative 0-8, 8-16, 16-24, 24-48 intervals
  Total amount of opioid delivered by the patient-controlled analgesia (PCA) device during the first 48 hours after surgery, recorded in milligrams (mg).

SECONDARY OUTCOMES:
QoR-15 Recovery Score | Postoperative 24th and 48th hours
  The investigators will use the Turkish version of Quality of Recovery (QoR) / QoR-15 questionairre
  PART A How have you been feeling in the last 24 hours? (0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent])
  Able to breathe easily Been able to enjoy food Feeling rested Have had a good sleep Able to look after personal toilet and hygiene unaided Able to communicate with Getting support from hospital doctors and nurses Able to return to work or usual home activities Feeling comfortable and in control Having a feeling of general well-being
  PART B Have you had any of the following in the last 24 hours? (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor]) Moderate pain Severe pain Nausea or vomiting Feeling worried or anxious Feeling sad or depressed
Dynamic and static Numeric Rating Scale scores | 0, 2, 4, 8, 16, 24, and 48 hours postoperatively
  Numeric Rating Scale (NRS) (0-10; 0= no pain, 10 = the most severe pain felt) pain scores at rest or movement at predefined postoperative hours
Total rescue analgesic dose | Postoperative 48 hours
  Despite the use of patient-controlled analgesia (PCA), if the Numeric Rating Scale (NRS) score is ≥4 at any time point, 0.5 mg/kg intravenous meperidine will be administered as rescue analgesia.
  Total amount of meperidin during the first 24 and 48 hours after surgery, recorded in milligrams (mg).
Time of first request for rescue analgesia | Postoperative 48 hours
  Despite the use of patient-controlled analgesia (PCA), if the Numeric Rating Scale (NRS) score is ≥4 at any time point, 0.5 mg/kg intravenous meperidine will be administered as rescue analgesia.
Length of Hospital Stay | Patients will remain under observation for at least 2 weeks until their postoperative discharge. Follow-up will be completed upon discharge. The length of hospital stay will be recorded.
  Length of hospital stay will be defined as the number of days from the end of surgery to hospital discharge
Block and Opioid-Related Adverse Effects and Complications | Postoperative 48 hours
  Block- and opioid-related adverse effects and complications, including but not limited to local anesthetic toxicity, hematoma, infection, nerve injury, nausea, vomiting, pruritus, sedation, and respiratory depression, will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Nilufer, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Girit M, Akin T, Narayanan M, Alici HA. Ultrasound guided quadro-iliac plane block: another novel fascial plane block. Pain Med. 2024 May 3;25(6):370-373. doi: 10.1093/pm/pnae018. PMID 38459608
- [Result] Turan EI, Sahin AS. Quadro-iliac plane block (QIPB) in lumbar stabilisation surgeries: A case series. Indian J Anaesth. 2025 Feb;69(2):244-245. doi: 10.4103/ija.ija_1077_24. Epub 2025 Jan 29. No abstract available. PMID 40160919
- [Result] Ciftci B, Ekinci M. A prospective and randomized trial comparing modified and classical techniques of ultrasound-guided thoracolumbar interfascial plane block. Agri. 2020 Nov;32(4):186-192. doi: 10.14744/agri.2020.72325. PMID 33398870